CLINICAL TRIAL: NCT06696937
Title: Comparative Effects of Tai Chi Vs Full Body Vibrator on Stress, Dynamic Balance, and Co-ordination Among Athletics Players.
Brief Title: Comparative Effects of Tai Chi vs Full Body Vibrator Among Athletic Players
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR and AHS/24/0415
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Sports Physical Therapy
Keywords: Tai chi,dynamic balance; Full body vibrator
MeSH Terms: interventions — Tai Ji

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tai chi (Experimental): Tai chi is a practice that involves a series of slow gentle movements and physical postures, a meditative state of mind, and controlled breathing. Tai chi originated as an ancient martial art in China. Over the years, it has become more focused on health promotion and rehabilitation.
  Interventions: Other: Tai chi
- Full body vibrator (Experimental): Advocates say that as little as 15 minutes a day of whole-body vibration three times a week may aid weight loss, burn fat, improve flexibility, enhance blood flow, reduce muscle soreness after exercise, build strength and decrease the stress hormone cortisol.
  Interventions: Other: full body vibrator

INTERVENTIONS:
Other: Tai chi — Tai chi is a practice that involves a series of slow gentle movements and physical postures, a meditative state of mind, and controlled breathing. Tai chi originated as an ancient martial art in China. Over the years, it has become more focused on health promotion and rehabilitation.
  Arms: Tai chi
Other: full body vibrator — Advocates say that as little as 15 minutes a day of whole-body vibration three times a week may aid weight loss, burn fat, improve flexibility, enhance blood flow, reduce muscle soreness after exercise, build strength and decrease the stress hormone cortisol.
  Arms: Full body vibrator

SUMMARY:
The aim of this study is to find out the Comparative effects of Tai chi and dynamic stretching exercises in reducing stress and insomnia among ameature athletics player's.

DETAILED DESCRIPTION:
In previous researches, little literature is available regarding comparison of the effectiveness of tai chi on insomnia and static balance among players.There is a dire need to explore the comparative effects of Tai chi and dynamic stretching exercises in reducing stress and insomnia among ameature athletics player's.

ELIGIBILITY:
Inclusion criteria:

* Female
* 17-35 years age
* Players with 2-3 years of experience in sports
* Minimum sports activity 1 hour 4 times a week

Exclusion criteria:

* Recreational players
* Players with recent injuries in the past 6 months
* Any neurological problem
* Player addicted to any drug or alcohol will be excluded

Ages: 17 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Female
Enrollment: 43 (Actual)
Dates: Start 2024-04-24 (Actual); Primary Completion 2024-11-20 (Estimated); Study Completion 2024-12-10 (Estimated)

PRIMARY OUTCOMES:
Modified bass test | 6 weeks
  The Modified Bass Balance Test is a clinical method for the assessment of functional jump-landing balance performance

CONTACTS AND LOCATIONS:
Overall Officials: Malia younas dr malia younas, pp-dpt, Principal Investigator — Riphah International University; Mishmal ammer Dr mishmal ammer, Dpt, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Pakistan Sports Academy, Lahore, Punjab Province
  - Pakistan Sports Board, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coughlan GF, Fullam K, Delahunt E, Gissane C, Caulfield BM. A comparison between performance on selected directions of the star excursion balance test and the Y balance test. J Athl Train. 2012 Jul-Aug;47(4):366-71. doi: 10.4085/1062-6050-47.4.03. PMID 22889651
- [Background] Nielsen MG, Ornbol E, Vestergaard M, Bech P, Larsen FB, Lasgaard M, Christensen KS. The construct validity of the Perceived Stress Scale. J Psychosom Res. 2016 May;84:22-30. doi: 10.1016/j.jpsychores.2016.03.009. Epub 2016 Mar 16. PMID 27095155
- [Background] Bai X, Xiao W, Soh KG, Agudamu, Zhang Y. 12-week concurrent brisk walking and Taijiquan (Tai Chi) improve balance, flexibility, and muscular strength of Chinese older women. PLoS One. 2023 Oct 26;18(10):e0293483. doi: 10.1371/journal.pone.0293483. eCollection 2023. PMID 37883372
- [Background] Huang HW, Nicholson N, Thomas S. Impact of Tai Chi Exercise on Balance Disorders: A Systematic Review. Am J Audiol. 2019 Jun 10;28(2):391-404. doi: 10.1044/2018_AJA-18-0115. Epub 2019 May 2. PMID 31046404
- [Background] Khuzema A, Brammatha A, Arul Selvan V. Effect of home-based Tai Chi, Yoga or conventional balance exercise on functional balance and mobility among persons with idiopathic Parkinson's disease: An experimental study. Hong Kong Physiother J. 2020 Jun;40(1):39-49. doi: 10.1142/S1013702520500055. Epub 2020 Feb 20. PMID 32489239
- [Background] Zhao J, Han W, Tang H. Lower limbs inter-joint coordination and variability during typical Tai Chi movement in older female adults. Front Physiol. 2023 May 2;14:1164923. doi: 10.3389/fphys.2023.1164923. eCollection 2023. PMID 37200836
- [Background] Wang C, Schmid CH, Fielding RA, Harvey WF, Reid KF, Price LL, Driban JB, Kalish R, Rones R, McAlindon T. Effect of tai chi versus aerobic exercise for fibromyalgia: comparative effectiveness randomized controlled trial. BMJ. 2018 Mar 21;360:k851. doi: 10.1136/bmj.k851. PMID 29563100
- [Background] Maciaszek J, Osinski W. The effects of Tai Chi on body balance in elderly people--a review of studies from the early 21st century. Am J Chin Med. 2010;38(2):219-29. doi: 10.1142/S0192415X10007798. PMID 20387220